CLINICAL TRIAL: NCT01965847
Title: Evening Dosing of Antihypertensive Medications in Chronic Kidney Disease Patients - A Pilot Study
Brief Title: Morning Versus Evening Dosing of Antihypertensive Medications: A Pilot Study to Assess Feasibility and Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UMNDrawz1
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Medication Therapy Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM dosing (Active Comparator): The study student pharmacist will perform medication therapy management with a focus on antihypertensive medications and specifically on the once daily antihypertensive assigned to MORNING dosing. Medication therapy management will take place in the clinic or by phone. Medication therapy management will include review of antihypertensive medications, patient empowerment and education, and provision of a personal medication record to the participant with specific instructions regarding the once daily antihypertensive medication assigned to morning versus evening. If a patient is taking more than one antihypertensive medication, only one will be used for the current study.
  Interventions: Behavioral: Medication therapy management
- PM dosing (Experimental): The study student pharmacist will perform medication therapy management with a focus on antihypertensive medications and specifically on the once daily antihypertensive assigned to EVENING dosing. Medication therapy management will take place in the clinic or by phone. Medication therapy management will include review of antihypertensive medications, patient empowerment and education, and provision of a personal medication record to the participant with specific instructions regarding the once daily antihypertensive medication assigned to morning versus evening. If a patient is taking more than one antihypertensive medication, only one will be used for the current study.
  Interventions: Behavioral: Medication therapy management

INTERVENTIONS:
Behavioral: Medication therapy management

SUMMARY:
Hypertension is a major risk factor for cardiovascular and renal disease, and a leading cause of premature mortality worldwide. Ambulatory blood pressure (BP) monitoring (ABPM) allows for assessment of BP throughout the day and night. Of all the BP measurements, nighttime systolic BP appears to be the best predictor of cardiovascular disease and all-cause mortality. Importantly, elevated nighttime BP is a modifiable risk factor; evening dosing of antihypertensive medications lower nighttime BP and reduces proteinuria. In a large, randomized controlled trial, evening dosing of antihypertensive medications reduced the hazard rate for major cardiovascular events by 67%. Findings were similar in the subgroup of participants with chronic kidney disease (CKD). However, this single-center study was designed to evaluate cardiovascular outcomes, not progression of CKD. The long-term effect of nighttime dosing of antihypertensive medications on progression of CKD is unknown.

To address this important gap in knowledge, the investigators plan to conduct a pragmatic, randomized controlled trial. 3600 participants at risk for progression of CKD who are taking ≥1 antihypertensive medication once daily will be randomized to morning versus evening dosing of at least one antihypertensive medication. The purpose of the current study is to obtain pilot data demonstrating the feasibility of the trial and the efficacy of the intervention.

DETAILED DESCRIPTION:
Background Hypertension is a major risk factor for cardiovascular and renal disease, and a leading cause of premature mortality worldwide. Early hypertension studies showed that treating elevated blood pressure (BP) reduces patients' risk of cardiovascular disease and all-cause mortality. In subsequent research, patients achieved greater improvement in cardiovascular outcomes when their treatment was aimed at a moderate systolic BP target (<150mmHg) than at higher targets. Although observational data suggest that even lower BP targets may be beneficial, this has not been seen in randomized trials; instead, "intense" treatment of hypertension (i.e., to a target systolic BP <120mmHg) was found to have no effect on participants' risk for renal disease, cardiovascular disease, or all-cause mortality. Similarly negative findings were reported in studies that enrolled participants with chronic kidney disease (CKD) and diabetes; all failed to demonstrate a benefit to intensive lowering of clinic BP.

One potential explanation for this apparent lack of benefit of intense BP targets is that the study protocols targeted reductions in clinic BP rather than ambulatory BP. Ambulatory BP monitoring (ABPM) allows for assessment of BP throughout the day and night. Of all the BP measurements, nighttime systolic BP appears to be the best predictor of cardiovascular disease and all-cause mortality. In fact, in most observational studies, clinic BP is no longer a predictor of adverse events after adjusting for nighttime BP. Importantly, elevated nighttime BP is a modifiable risk factor; evening dosing of antihypertensive medications lower nighttime BP and reduces proteinuria. In a large, randomized controlled trial, evening dosing of antihypertensive medications reduced the hazard rate for major cardiovascular events by 67%. Findings were similar in the subgroup of participants with CKD. However, this single-center study was designed to evaluate cardiovascular outcomes, not progression of CKD. The long-term effect of nighttime dosing of antihypertensive medications on progression of CKD is unknown.

To address this important gap in knowledge, the investigators plan to conduct a pragmatic, randomized controlled trial. 3600 participants at risk for progression of CKD who are taking ≥1 antihypertensive medication once daily will be randomized to morning versus evening dosing of at least one antihypertensive medication. The purpose of the proposed study is to obtain pilot data demonstrating the feasibility of the trial and the efficacy of the intervention.

Overview of Trial Design The study will be conducted in the renal clinic at University of Minnesota Medical Center (UMMC). Eligible patients will have chronic kidney disease and be taking a once daily antihypertensive medication. Participants will be randomized to receive their once daily antihypertensive medication in the morning or the evening. Medication therapy management with a focus on antihypertensive medications will take place at the time of a clinic visit or via phone after the clinic visit. Adherence to medications will be assessed 3-6 weeks after the clinic visit.

Objective The primary objective of this pilot study is to demonstrate 1) the feasibility of a simple randomized trial and 2) the efficacy of medication therapy management for assigning participants to take a once daily antihypertensive medication either in the morning or in the evening.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe kidney disease, defined as:

   1. Estimated glomerular filtration rate 20-45 mls/min/1.73m2; or
   2. Estimated glomerular filtration rate: 45-60 mls/min/1.73m2 with proteinuria defined by either a urine albumin to creatinine ratio >300mg/g or a urine protein to creatinine ratio >500mg/g.
2. Age 19-80 years
3. Taking one or more non-diuretic antihypertensive medication once daily
4. Appointment at the University of Minnesota Medical Center Renal Clinic.

Exclusion Criteria:

1. Pregnant women
2. Patients that are difficult to follow-up with: prisoners, non-English speakers
3. Patients with adherence difficulty: Mentally disabled, emotionally disabled, developmentally disabled, impaired decision making capacity.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04-17 (Actual); Study Completion 2015-04-17 (Actual)

PRIMARY OUTCOMES:
Adherence to timing instructions | 3-6 weeks after intervention
  Participants will be called three to six weeks after their clinic visit by study personnel. Participants will be asked the following questions about the once a day antihypertensive medication involved in the study: "In the last seven days, how many times did you take [name of antihypertensive medication] in the morning? In the last seven days, how many times did you take [name of antihypertensive medication] in the evening?"

SECONDARY OUTCOMES:
General medication adherence | 3-6 weeks after intervention
  Participants will be called three to six weeks after their clinic visit by study personnel. Participants will be asked about general medication adherence using the Morisky medication scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Smith JR, Hillman L, Drawz PE. Pharmacist-based antihypertensive medication review and assignment of morning versus evening dosing of once-daily antihypertensive medications: A pilot study to assess feasibility and efficacy in chronic kidney disease patients. Clin Exp Hypertens. 2018;40(6):569-573. doi: 10.1080/10641963.2017.1411493. Epub 2017 Dec 6. PMID 29211509